CLINICAL TRIAL: NCT06371066
Title: The Effect of Video-based Training on the Knowledge Levels of Nursing Students: A Randomized Controlled Trial
Brief Title: The Effect of Video-based Training on the Knowledge Levels of Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Elif Akyüz, Associate professor, Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EAkyuz-2
Record Dates: First submitted 2024-04-09; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Student Nursing; Medical-surgical Nursing; Nursing Care; Education
Keywords: Nursing students; video-based training; preoperative education; preoperative preparation
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: intervention, control
Who Masked: Outcomes Assessor
Masking Description: it was an educational intervention. All participants were in the same class so we blinded only statisticians.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): video-based training group
  Interventions: Other: experimental group
- Control group (Other): traditional formal training group
  Interventions: Other: Control group

INTERVENTIONS:
Other: experimental group — the experimental group was educated by video
  Other Names: video based education
  Arms: Experimental group
Other: Control group — the control group was educated by traditional formal training
  Other Names: tradional formal education
  Arms: Control group

SUMMARY:
Although face-to-face education is widely used as a traditional method, emerging computer technology has allowed new training approaches such as video-based training (VBT) platforms to flourish, especially in the last four decades. Educators adopted VBT as a cost-effective and accessible medium to address some of their training needs. It contains purposely designed visual cues and draws learners' attention during the learning process, and the dynamic details enable learners to better understand the learning contents. The use of new technologies such as e-learning, computer-assisted learning, VBT, and web-based applications for clinical skill education has increased learner satisfaction compared with conventional education methods. Preoperative patient preparation is a crucial element of preoperative nursing care. A surgical nurse is a specialized coordinator of patient care, and the main purposes of this role are to meet the patient's and the family's needs individually and to prepare them for the scheduled procedure and postoperative recovery. Preoperative patient preparation contains multiple components and steps such as preoperative education, including physical, social, psychological, and legal preparation, and preparation for the night and day of surgery. the nature of the process has many components and steps, it is not easy for students to learn this subject, and nursing educators were able to experience this in a clinical practice environment. And the educators started to search for new teaching techniques to teach this subject like the other colleagues. the investigator's aim in this project is to determine the effect of VBT on the knowledge levels of nursing students on preoperative patient preparation when compared to traditional training methods.

DETAILED DESCRIPTION:
This pretest-posttest randomized controlled experimental study was designed as a randomized controlled parallel designed trial.

This study was conducted at the nursing department of a state university. The population of the study consisted of second-year nursing students who enrolled in the Surgical Nursing course. The study was conducted with students who met the inclusion criteria in the study without any sample calculation. Class size was 100 and 97 of them agreed to participate in the study. The students were assigned to the VBT group or the traditional training group via a stratified randomization method in order to ensure the balance between the groups. The study was carried out with 49 experimental and 48 control groups. After the students were divided into two groups according to gender, an equal number of male and female students were assigned to the experimental and control groups by drawing lots, one of the simple random sampling methods. The student participants were randomly assigned to one of the two groups using a random number table. To avoid bias in this randomized controlled study, assignments to the groups were made by an outside researcher. All training sessions were carried out by researchers. Dependent variables of the research project are; students' level of knowledge, and the independent variables are student information data. Data collection forms (student information, knowledge levels) developed by researchers using the literature

Video scenario: It consisted of a preoperative patient case, learning objectives for nursing care, the content of the scenario and the roles. The scenario involved one 65-year-old female patient who had weight loss, loss of appetite, abdominal pain, and bloating for preoperative preparation of left hemicolectomy surgery. It has been prepared by the formal education given within the scope of the surgical nursing course. The scenario was designed with careful consideration given to conceptual, psychological, and physical realities. The content validity of scenario was assessed by four expert nursing faculty members.

İmplementation: The training was presented to the experimental group by video, and to the control group by the traditional method (using a lecture-style PowerPoint presentation with supporting visual components, question-answer, and narrative method). Before the training, both groups answered the "The Student Information Form" and "The Knowledge Form" and were informed about the purpose of the course, learning objectives and outcomes, and scenario roles, and their questions were answered. The students were informed that their involvement in the research was voluntary and had no bearing on their course grades no academic credit would be given for participating. At the end of the training of both groups, all the scenario was discussed with the students, and their questions were answered. Right after training (post-test 1) and three weeks later (post-test 2: two weeks after post-test 1), the students answered 'The Knowledge Form'.

ELIGIBILITY:
Inclusion Criteria:

* willingness to participate in the study,
* taking no previous surgical nursing course.

Exclusion Criteria:

* unwillingness to participate in the study
* having no previous knowledge and experience in surgical nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
The Student Information Form | one day
  This form was developed by the researchers in accordance with the literature. It consisted of 12 questions about individual (age, gender, economic status), academic (graduated high school), and experiencing video in daily life (taking VBT before, status and frequency of watching training videos on the internet) characteristics.
The Knowledge Form for Preoperative Patient Preparation | one day
  This form was prepared by the researchers in line with the literature. The form consisted of 25 items with three options (True, False, Not know). Each right answer was given one points, while each wrong and not known answer was given zero points. The total test score ranged from zero to 25. High scores indicated a high level of knowledge. In order to evaluate whether it looked or read like the construct aiming to measure the level of knowledge of preoperative education and patient preparation on the day of surgery was assessed by four expert nursing faculty members. The form was revised and finalized in line with expert evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Atiye Erbas, PhD, Principal Investigator — Duzce University
Locations (1):
- Kirikkale University, Kırıkkale, Turkey (Türkiye)